CLINICAL TRIAL: NCT02590835
Title: Efficiency of Piezocision-assisted Orthodontic Treatment in Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. France LAMBERT (Other)
Responsible Party: Sponsor-Investigator, Dr. France LAMBERT, Professor, University of Liege
Organization: University of Liege (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2013-3
Record Dates: First submitted 2015-10-21; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Tooth Overcrowding
Keywords: Adult patients; Patient demand for orthodontic treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Treated with conventional orthodontics
  Interventions: Procedure: Orthodontic procedures (for both groups : Control group and Test group)
- Test group (Experimental): subjected to piezo-assisted orthodontics
  Interventions: Procedure: Orthodontic procedures (for both groups : Control group and Test group); Procedure: Piezo-assisted orthodontics (only the Test group)

INTERVENTIONS:
Procedure: Orthodontic procedures (for both groups : Control group and Test group) — Damon self-ligating systems (Ormco, Orange, Calif) were used for all patients. The patients were allowed to choose between clear or metal brackets. The bonding method was standardized and applied according to the manufacturer's instructions. After bracket bonding, 0.014-in copper-nickel-titanium Damon arch forms were placed. The subjects were recalled every two weeks, and the archwires were changed only when full bracket engagement was achieved. The sequence of archwires was as follows: 0.018-in, 0.014x0.025-in and 0.018x0.025-in copper nickel-titanium archwires for alignment; and 0.019x0.025-in stainless steel archwires for fine-tuning. Following the alignment steps, impressions were taken, and blinded orthodontic consultants validated appliance removal or provided advice regarding further adjustments. Alginate impressions were taken after the removal of the appliances, and both fixed and removable retainers were placed.
Procedure: Piezo-assisted orthodontics (only the Test group) — The piezocisionTM surgery was performed one week after orthodontic appliance placement . The patients received local anesthesia in both arches, and vertical interproximal micro-incisions were created below each interdental papilla. In cases of root proximity (i.e., less than 2 mm of interdental bone), this procedure was not applied. These incisions were kept to a minimum (varying from 5 mm to 8 mm). Next, using a vertical piezoelectric device, 5-mm long and 3-mm deep corticotomies were made, and no subsequent sutures were required needed (figure 1). The patients were advised to take analgesics (paracetamol) only if necessary and to record their daily intakes for one week. Anti-inflammatories were prohibited to avoid interference with the RAP. Careful tooth brushing and the use of a mouthwash (chlorhexidine 0.2% Perio-Aid, Dentaid Benelux, Houten, Netherlands) were recommended for 7 days.
  Arms: Test group

SUMMARY:
This study was designed as a randomized controlled clinical trial to compare conventional orthodontic treatment (control group) and piezocision-assisted orthodontic treatment (PS group). Twenty-four consecutive adult patients from the Orthodontics Department of Liege University Hospital, Belgium who met the inclusion criteria were enrolled from January to October of 2013.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (completed growth)
* Maxillary and mandibular overcrowding
* Patient demand for orthodontic treatment
* Adequate dento-oral health
* ASA I and ASA II
* Compliance with clinic visits every 2 weeks

Exclusion Criteria:

* A need for tooth extraction
* A need for orthodontic temporary anchorage devices
* A history of periodontal disease
* Smokers
* Altered bone metabolism (e.g., due to anti-resorptive drug, steroid or immunosuppressant use)
* Mental or motor disabilities
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Overall treatment time measurement (in days) | 3 years
  Comparaison of the overall treatment time between the test group (piezocision group) and the control group will be performed. It will be evaluated by measuring the time (in days) between the placement and the debond of the orthodontic appliance. The hypothesis is that piezocision accelerate orthodontic tooth movement.

SECONDARY OUTCOMES:
Root resorption parameters measurements (intrabuccal radiographic in millimeters) | 3 years
  A comparaison of orthodontic parameters (root resorption) between the test group and the control group before and after orthodontic treatment will be performed. The root resorption will be measured in intrabuccal radiographic (millimeters) on the day of the placement of this appliance and at the debond.
Comparaison of periodontal parameters between the test group and the control group before (at baseline) and after orthodontic treatment. | 3 years
Patient-centered outcomes (VAS questionnaire) | 7 days
  Satisfaction post treatment using a VAS questionnaire and analgesic consumption (milligrams of paracetamol) during 7 days after the placement of the orthodontic appliance.

REFERENCES:
- [Derived] Charavet C, Lecloux G, Bruwier A, Rompen E, Maes N, Limme M, Lambert F. Localized Piezoelectric Alveolar Decortication for Orthodontic Treatment in Adults: A Randomized Controlled Trial. J Dent Res. 2016 Aug;95(9):1003-9. doi: 10.1177/0022034516645066. Epub 2016 Apr 29. PMID 27129491